CLINICAL TRIAL: NCT04827563
Title: Risk Factors for Dyspnea and Cardiotoxicity in Patients With Multiple Myeloma Who Receive Carfilzomib: A Prospective Pilot Study
Brief Title: Dyspnea and Cardiotoxicity in Multiple Myeloma Patients Who Receive Carfilzomib
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-1768
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Shortness of Breath; Dyspnea; Cardiotoxicity
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Dyspnea; Cardiotoxicity | interventions — Echocardiography; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with Normal Baseline Endothelial Function
  Interventions: Device: EndoPAT; Device: Blood Pressure Cuff; Diagnostic Test: Echocardiogram; Other: Quality of Life Assessment; Other: Blood Tests
- Participants with Abnormal Baseline Endothelial Function
  Interventions: Device: EndoPAT; Device: Blood Pressure Cuff; Diagnostic Test: Echocardiogram; Other: Quality of Life Assessment; Other: Blood Tests

INTERVENTIONS:
Device: EndoPAT — An FDA approved device to test the health of a patient's blood vessels, which involves putting an oxygen probe on the participant's finger.
Device: Blood Pressure Cuff — A device used to conduct blood pressure monitoring using a home blood pressure cuff that participant wears for 24 hours.
Diagnostic Test: Echocardiogram — A test used to conduct an ultrasound of participant's heart.
Other: Quality of Life Assessment — A survey that will be given to participants to report their quality of life and symptoms related to multiple myeloma.
Other: Blood Tests — Routinely collected for all participants who begin carfilzomib treatment.

SUMMARY:
This study will explore why some multiple myeloma patients who receive carfilzomib (an anti-cancer medication) experience shortness of breath while others do not. The purpose of this research is to gather information on the effectiveness of the EndoPAT device, which is FDA-approved to assess the health of a patient's blood vessels. These assessments will help doctors leading the study determine the reasons why patients may develop shortness of breath (dyspnea) when being treated with carfilzomib and ways to better prevent this shortness of breath.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmed diagnosis of multiple myeloma
* Newly-diagnosed multiple myeloma, or relapsed/refractory multiple myeloma with receipt of 1-3 previous lines of therapy and with a 2-week washout from prior therapy
* Receiving carfilzomib as either standard-of-care therapy or as part of a clinical trial

Exclusion Criteria:

* Previous receipt of anthracycline chemotherapy
* Previous receipt of carfilzomib
* Four or more previous lines of therapy
* Active pregnancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with multiple myeloma who are being treated with carfilzomib.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function and Dyspnea Associations in Multiple Myeloma Patients | 2 months
  The association between baseline endothelial function and dyspnea in myeloma patients treated with carfilzomib. These associations will be assessed by comparing endothelial function within two cohorts: patients with abnormal baseline endothelial function, and patients with normal baseline endothelial function. Baseline endothelial function will be measured using EndoPat, an FDA-approved device used for health tests. Dyspnea rates will be assessed by participant-reported outcomes using the FACIT Dyspnea-10 Raw Dyspnea Score and Common Terminology Criteria for Adverse Events V5.

SECONDARY OUTCOMES:
Cardiovascular Toxicities Associated with Changes in Carfilzomib-Induced Endothelial Function | 2 months
  The association between changes in carfilzomib-induced endothelial function and frequency of cardiovascular toxicities stratified by patients with abnormal and normal baseline endothelial function.Cardiovascular toxicities in this study will be defined as new or worsening symptomatic heart failure, hypertension, myocardial ischemia, stroke, pulmonary hypertension, arrhythmias and thromboembolic events that will be measured per CTCAE V5.
The Affects of Carfilzomib Dose/Dosing Schedule on the Incidence of Dyspnea | 2 months
  The affects of carfilzomib dose/dosing schedule on how often participants experience dyspnea (shortness of breath) will be assessed by participant reported outcomes using the FACIT Dyspnea-10 (raw dyspnea score) and data collected on adverse events (side effects) using CTCAE V5.
Changes in Cardiovascular Physiology and Risk Factors Associated with Endothelial Function | 2 months
  To determine whether changes in endothelial function are associated with cardiovascular physiological changes and cardiovascular risk factors within participants receiving carfilzomib. These associations will be measured by: hemodynamics (using the average 24-hour ambulatory blood pressure reported by participants after treatment using home blood pressure monitoring), echocardiography using echocardiogram, and data collected on patient's vascular and cardiovascular health at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne DeCara, MD, Principal Investigator — University of Chicago - Comprehensive Cancer Center
Locations (1):
- University of Chicago, Chicago, Illinois, United States